CLINICAL TRIAL: NCT05747781
Title: Validation of Standardized Tests Allowing the Evaluation of the Impacts of Glaucomatous Optic Neuropathy in Daily Life Activities
Brief Title: STReetlab Assessment Tool of Activities Daily Living in Glaucoma Patient
Acronym: STRATAL-GL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P22-05; 2022-A02573-40 (Registry Identifier: IDRCB-ANSM)
Record Dates: First submitted 2023-02-02; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Optic Neuropathy
MeSH Terms: conditions — Optic Nerve Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, longitudinal, non-randomized, open-label study with glaucoma patients and control group (healthy volunteers)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilot Phase (Active Comparator): 12 patients with glaumatous optic neuropathy
  Interventions: Behavioral: Pilot Phase: standardized behavioral task
- Validation Phase (Placebo Comparator): 66 patients with glaumatous optic neuropathy 12 subjects with no known visual impairment
  Interventions: Behavioral: Validation Phase: standardized behavioral task

INTERVENTIONS:
Behavioral: Pilot Phase: standardized behavioral task — Pilot Phase:
  * Mobility under variable light conditions (scotopic, photopic, glare, dark adaptation), performed in a virtual environment.
  * Visual search for objects in real life scenes (office, kitchen, living room) performed in a virtual environment.
  * Ability to drive (UFOV and DVFAT psychophysical tests).
  Arms: Pilot Phase
Behavioral: Validation Phase: standardized behavioral task — Validation Phase:
  * Mobility in variable light conditions (photopic and scotopic), performed in real and virtual environments.
  * Visual search for objects in real scenes (office, kitchen, bedroom, living room) performed in a virtual environment.
  * Driving ability (two psychophysical tests UFOV and DVFAT, one supervised road test).
  Arms: Validation Phase

SUMMARY:
The impact of glaucomatous optic neuropathy on the daily life of patients is poorly characterized and does not benefit from standardized tests.

The development and validation of new tests could be used to assess the efficacy of innovative treatments for visually impaired patients and/or optimize management strategies.

DETAILED DESCRIPTION:
This study will be conducted with 2 groups of subjects: glaucoma patients and healthy volunteers.

The objective of this project is to validate performance criteria (PerfO) using standardized tasks to assess the quality of life of patients but also to better judge the severity of glaucoma damage. The fidelity, reproducibility, validity and sensitivity of these new tests will be studied. This study will include two phases: a pilot phase to refine the parameters of the tests for the target population, and a validation phase for the tools.

This study will be performed in two phases: pilot phase and validation phase.

Pilot phase (12 months): 12 glaucoma patients (4 stage 1; 4 stage 2 and 4 stage 3), the objective of this phase is to define the optimal parameters of task content, as well as the conditions of luminosity and contrast.

Validation phase: 66 glaucoma patients classified into 3 groups of 22 patients according to the stage of severity (22 stage 1; 22 stage 2 and 22 stage 3) and 22 healthy volunteers matched for age and sex (matching rules ± 5 years).

The objective of this phase is to validate tests that will allow the evaluation of the impact of peripheral visual impairment on the sensory and motor performances of patients in their daily life.

ELIGIBILITY:
Inclusion Criteria:

Glaucoma patients:

* Age: 18 - 80 years,
* Visual acuity of at least 6/10th binocular,
* Patient followed at Quinze-Vingts and presenting with chronic stable glaucoma defined by the glaucoma ophthalmologist,
* MMSE questionnaire score ≥ 25/30 or ≥ 16/25 (if the patient no longer drives),
* Ability to give consent and comply with the study protocol,
* Person with Social Security coverage.
* Recruitment of glaucoma patients will be based on the criteria defined by the HPA classification (Appendix) on the basis of the Humphrey visual field, for categorization of patients into three stages of optic neuropathy progression (early stage "1", moderate "2" and advanced "3").

For the optional roadside fitness visit (V4), specific inclusion criteria will be required for this study: the roadside assessment will be performed with volunteers (GL and VS) who report being:

* Always drivers in possession of a valid driver's license,
* Driven at least 500 km in the past year.

Healthy volunteer:

* Age: 18 - 80 years.
* Age and sex matching between healthy volunteers and glaucoma patients (± 5 years).
* MMSE questionnaire score ≥ 25/30.
* Visual acuity of at least 10/10th in binocular.
* Ability to give consent and comply with the study protocol.
* Person with a Social Security plan.

For the roadside fitness visit (V4), specific inclusion criteria will be required for this study: the roadside assessment will be performed with volunteers who declare themselves:

* Always drivers in possession of a valid driver's license,
* Driven at least 500 km in the past year.

Exclusion Criteria:

* Pregnant women.
* Inability to personally give consent.
* Participants will not have neurodegenerative diseases or any other disease that could interfere with the assessments planned during this study.
* Participants will not have any other ophthalmologic diseases other than glaucoma.
* Drug treatments that may cause motor, visual, or cognitive impairment (PSAs, neuroleptics, etc.) or that may interfere with the study assessments.
* Condition that limits ability to move.
* Inability to read.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Discrimination capacity | 6 months
  Number of patients with capacity of discrimintaion compared to healthy volunteers
Reproducibility of performance tests | 6 months
  Number of patients able to reproduce the same performance tests
Analysis reationships between Performance Outcomes (PerfO), Patient-ReportedOutcome (PRO) and Clinical Outcomes. | 6 months
  Number of patients in each situation

SECONDARY OUTCOMES:
Postural control | 6 months
  Number of patients with modification of Romberg quotient to assess whether the central nervous system has re-weighted the weight of visual, vestibular and proprioceptive inputs with the onset of glaucomatous optic neuropathy.
Oculomotricity: | 6 months
  Number of patients with alteration of eye movement parameters during fixation tasks, ocular tracking (number of fixations, fixation error (gain), speed and number of catch-up saccades) and saccades) and ocular saccades.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe BAUDOUIN, Pr, Principal Investigator — Hôpital National de la Vision des15-20